CLINICAL TRIAL: NCT03260218
Title: Protocol for a Single-Centre Prospective Observational Study of Postoperative Delirium Following Total Joint Arthroplasties Among South East Asians
Brief Title: Protocol for Observational Study of Post op Delirium Following Total Joint Arthroplasties
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJA2017
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; elderly; total joint replacement; risk factors for delirium; postoperative confusion
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of post-operative delirium in the South-east Asian population is not known. Through a prospective, single centre, observational study, the investigators aim to characterize the incidence and risk factors of delirium in older adults undergoing elective total joint arthroplasties (TJA). The study will recruit eligible patients (65 - 90 years old undergoing elective TJA), with a targeted sample size of 500. Patients will be screened for dementia and Confusion Assessment Method (CAM) scores obtained pre and post operatively. Other data such as preoperative Charlson comorbidity index (CCI), post op complications using Post operative Morbidity Survey (POMS), pain scores, readmission rates and length of hospital stay (LOS), functional and health-related quality-of-life (HRQoL) will also be collected and analysed.

DETAILED DESCRIPTION:
BACKGROUND

Modern studies have evaluated the risk factors and incidence of postoperative delirium in post-TJA patients. In current literature, incidence ranges from 0-10%. However, the epidemiology of these studies mainly focused on non-Asian populations. The investigators hope to determine both the incidence and risk factors of postoperative delirium in patients undergoing TJA with a focus on the Asian population. This is especially relevant in today's ageing Asian population.

AIMS

To characterize the incidence and risk factors of delirium in older adults undergoing elective total joint replacement surgery.

HYPOTHESIS

The incidence of postoperative delirium following elective TJA is low compared to Western studies. Age, gender and use of opioids perioperatively are risk factors for postoperative delirium following elective total joint replacement surgery.

DESIGN: Prospective observational study.

SETTING: Academic medical center.

DURATION: July 2017 - Dec 2017

STUDY POPULATION: Individuals aged 65 to 90 years old undergoing elective total joint (hip or knee) replacement surgery.

METHODOLOGY:

Preoperative data

Before the operation, each patient will be interviewed to assess their baseline cognitive status. The Mini-Mental State Examination (MMSE) will be used, which is a 11-question screening tool used to evaluate the cognitive aspects of mental function. A score of 0-30 can be obtained with higher values denoting better cognitive function. A score of <24 suggests cognitive impairment. A MMSE test modified for use in Singapore will be use, due to cultural and climate differences. In addition, the test will be administered in English, Chinese or Malay, according to the language the participant is most well-versed in. The Chinese and Malay versions of MMSE have similar test questions and are scored the same way as the English version. Sensory impairment will be assessed during the preoperative interviews. Patients will be asked to wear their visual or hearing aids during these interviews. A patient will be considered to have visual or hearing impairment if the research member conducting the interview is unable to perform the interview normally due to the sensory impairment, such as raising his/her voice for a patient with impaired hearing. The grip strength of each patient will also be measured using the JAMAR® Plus+ Digital Hand Dynamometer (Sammons Preston Inc, Bolingbrook, IL). The patient baseline characteristics will be obtained from the medical records. Perioperative data is available through the Preoperative Evaluation Clinic (PEC) database as well as the Orthopaedic Diagnostic Centre (ODC) total joint registry, which will be prospectively entered into the REDCap™ database. This will include data regarding patient's demographics, smoking history, alcohol history, pre-existing medical conditions, preoperative medications. Each patient will also be rated preoperatively by an anaesthesiologist in the PEC based on the American Society of Anaesthesiologists (ASA) physical status classification. For analysis, the investigators will be calculating each patient's perioperative risk based on the Charlson Comorbidity Index (CCI). Preoperative laboratory results, including data about haemoglobin or creatinine level, will also be collected.

Intraoperative data

Data regarding the surgery will be collected. Intraoperative data includes type of arthroplasty performed (total hip or total knee arthroplasty), type of anaesthesia (spinal, general or other anaesthesia), use of femoral nerve block, intraoperative drug use, tourniquet time, intra-articular injections and blood transfusion (number of pints transfused). Occurrence of hypotension, which is defined as a mean arterial pressure <60mmHg, and its duration will also be recorded.

Postoperative data

Primary outcome

The primary outcome will be the presence of postoperative delirium following TJA. Each patient will be assessed for delirium on postoperative day (POD) 1, 2 and 3 in the wards at 7am as well as the day of discharge. Delirium will not be evaluated on POD 0 due to difficulty in differentiating delirium from the effects of residual anaesthesia. The Confusion Assessment Method (CAM) will be used to detect postoperative delirium and delirium severity. Delirium is said to be present if the patient meets the CAM criteria for any of the postoperative assessments. Patients assessed to have delirium will be referred to the psychiatrists for further management.

Short-term secondary outcomes

Postoperative complications will be quantified by the Postoperative Morbidity Survey (POMS). This survey will be conducted on the day-of-discharge and there will be surveillance for up to 30 days following index surgery. Postoperative delirium and delirium severity will be assessed using CAM. Hospital-based outcomes will be obtained from the medical records. Perioperative data is available through the PEC database as well as the ODC total joint registry. All perioperative data and clinical outcomes will be analyzed. The incidence of postoperative delirium will be calculated using standard formula. Regression analysis will be performed to identify risk factors for delirium. The incidence of 30 day post operative complications will also be screened for and collected using the Post-operative Morbidity Survey (POMS), at the point of discharge and 30 days from date of surgery.

Long-term secondary outcomes

Longer-term outcomes such as functional and health-related quality-of-life (HRQoL) outcomes will also be recorded by the ODC total joint registry at 6 months, 1 year, 2 years and 5 years postoperatively. Knee function will be measured using the new Knee Society Knee Score (KSKS) and Function Score (KSFS)29. The KSKS and KSFS each range from 0 (worst) to 100 (best). In addition, the Oxford Knee Score (OKS)31 will also be used, which is a 12-item, patient-assessed questionnaire designed specifically for use in patients undergoing TKA. Each item is scored from 1 (least difficulty/severity) to 5 (most difficulty/severity), and individual item scores are summed to yield an overall score ranging from 12 (no pain or limitation) to 60 (severe pain or limitation). HRQoL will be assessed based on the 36-Item Short Form Health Survey (SF-36) to obtain a baseline score. It consists of 36 questions categorised into 8 domains (physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions). Higher scores indicate better health status and quality of life. Days alive and out of hospital (DAOH) will also be determined for each patient at 1 month, 6 months and 12 months to assess overall impact of postoperative delirium on morbidity and mortality. DAOH will be calculated based on death date (if present) and duration of all subsequent hospitalisations until the follow-up date. This will be recorded as a percentage by dividing DAOH by total potential follow-up period, which is the time period between the operation and the respective dates of follow-up (1 month, 6 months and 12 months).

Postoperative risk factors

Other postoperative data will be collected as variables for risk factors. Postoperative pain at rest will be evaluated using the pain Visual Analog Scale (VAS) during the same visit as CAM on POD 1, 2 and 3. Each patient will score pain experienced at rest on a scale, with 0 = no pain and 10 = maximum pain. Sensory impairment will also be assessed during the postoperative interviews similar to the preoperative assessments.

Data Management

Patient data will be kept confidential throughout the study. All electronic study data entry, storage and analysis will be done according to institutional data security policy, using password protected data in secure systems. The patient data collected will be de-identified and the key kept securely separated with access limited to principal investigator and co-investigators. A study-related identification number given to each patient will be used on the case report form. Research members will enter the de-identified data into the REDCap™ (Research Electronic Data Capture) tool hosted on a secure server at Singapore General Hospital. The hardcopy of the research data will be securely stored within the department. The softcopy of research data will be saved in a password-protected file and will be stored in institution approved login-protected system and encrypted hard-drive. Only study members will have access to the data.

Power and sample size calculations

The sample size will be calculated based on the incidence of postoperative delirium. Based on existing literature, the estimated incidence of postoperative delirium following TJA is around 10%. Using this estimate, a minimum sample size of 150 patients will be needed to detect the incidence with a precision of 5% and power of 80%. The sample size of 200 patients is needed to measure incidence to account for attrition.

However, this study will also be analysing the factors which may be correlated to postoperative delirium by logistic regression. A study population size of 500 will thus be targeted to be able to run a multiple logistic model while minimising the limitation of a small number of events of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective total knee or total hip arthroplasty

Exclusion Criteria:

* Patients who are deemed to lack mental capacity to give consent.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged between 65 and 90 undergoing elective total joint (hip or knee) replacement surgery in Singapore General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Post operative delirium incidence | Up to 30 days
  Measured using confusion assessment method (CAM) tool

SECONDARY OUTCOMES:
Post operative complications | Up to 30 days post operatively
  measured using post operative morbidity survey (POMS)
incidence of post operative nausea and vomiting (PONV) | post op day 1
  the total number of patients experiencing PONV
Length of hospital stay | up to 12 months
  the total number of days stayed in hospital during this elective admission
Hospital readmission rate | 30 days post operative
  the percentage of patients being readmitted for a complication related to the surgery
functional and health-related quality-of-life (HRQoL) | 6 months , 12 months
  tools used to assess knee function, ADL status, emotional and social wellbeing
Days Alive and Out of Hospital (DAOH) | 1 month, 6 months, 12 months
  measures the death rate and total summation of days spent outside of hospital following the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Abdullah HR, Tan SR, Lee SJ, Bin Abd Razak HR, Seet RH, Ying H, Sethi E, Sim EY. Protocol for a single-centre prospective observational study of postoperative delirium following total joint arthroplasties among South East Asians. BMJ Open. 2018 Mar 6;8(3):e019426. doi: 10.1136/bmjopen-2017-019426. PMID 29511014